CLINICAL TRIAL: NCT01630460
Title: Identification of Mutations That Lead to Craniometaphyseal Dysplasia in Families and Isolated Cases and Studies of Cellular and Molecular Mechanisms
Brief Title: Genetic and Functional Analysis of Craniometaphyseal Dysplasia (CMD)
Acronym: CMD
Status: Recruiting | Type: Observational
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Ernst Reichenberger, Assoc. Prof., UConn Health
Other Study IDs: UCHC03-008CMD
Record Dates: First submitted 2012-06-25; First posted 2012-06-28 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Craniometaphyseal Dysplasia
Keywords: Craniometaphyseal dysplasia; bone; hyperostosis; osteoblast; osteoclast
MeSH Terms: conditions — Schwartz-Lelek syndrome; Hyperostosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, blood, bone tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
CMD can be inherited in an autosomal dominant or recessive trait. CMD may also be caused by de novo mutations. The goal of this study is to identify genes and regulatory elements on chromosomes that are the cause for CMD. The investigators also study blood samples and tissue samples from patients to learn about the processes that lead to this disorder. The investigators long-term goal is to find mechanisms to slow down bone deposition in CMD patients.

DETAILED DESCRIPTION:
CMD is a very rare bone disorder that affects mostly bones of the head (=cranial bones) but also long (=tubular) bones. Therefore, CMD has been added to the class of craniotubular bone disorders. There are a number of disorders in this group and sometimes they are difficult to distinguish. Typical signs for CMD are the lifelong bone deposition in bones of the face and head (=progressive craniofacial hyperostosis) and the widening of the ends of long bones (=metaphyseal flaring). Typical facial characteristics are wide-set eyes and a prominent jaw (=mandible). CMD is sometimes diagnosed in infants. The best way to confirm diagnosis is by molecular genetics.

ELIGIBILITY:
Inclusion Criteria:

* CMD; unaffected individuals only if part of a participating CMD family

Exclusion Criteria:

* No CMD; unaffected individuals only as part of a participating CMD family

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with diagnosed CMD
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2009-04; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic elements | at time of identification
  The goal is to identify relevant genes or genetic elements that cause the disease or contribute to the disease progression and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ernst J Reichenberger, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Result] Dutra EH, Chen IP, McGregor TL, Ranells JD, Reichenberger EJ. Two novel large ANKH deletion mutations in sporadic cases with craniometaphyseal dysplasia. Clin Genet. 2012 Jan;81(1):93-5. doi: 10.1111/j.1399-0004.2011.01700.x. No abstract available. PMID 22150416
- [Result] Chen IP, Wang L, Jiang X, Aguila HL, Reichenberger EJ. A Phe377del mutation in ANK leads to impaired osteoblastogenesis and osteoclastogenesis in a mouse model for craniometaphyseal dysplasia (CMD). Hum Mol Genet. 2011 Mar 1;20(5):948-61. doi: 10.1093/hmg/ddq541. Epub 2010 Dec 13. PMID 21149338
- [Result] Chen IP, Wang CJ, Strecker S, Koczon-Jaremko B, Boskey A, Reichenberger EJ. Introduction of a Phe377del mutation in ANK creates a mouse model for craniometaphyseal dysplasia. J Bone Miner Res. 2009 Jul;24(7):1206-15. doi: 10.1359/jbmr.090218. PMID 19257826
- [Result] Reichenberger E, Chen IP. Autosomal Dominant Craniometaphyseal Dysplasia. 2007 Aug 27 [updated 2025 Aug 14]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1461/ PMID 20301634
- [Result] Reichenberger E, Tiziani V, Watanabe S, Park L, Ueki Y, Santanna C, Baur ST, Shiang R, Grange DK, Beighton P, Gardner J, Hamersma H, Sellars S, Ramesar R, Lidral AC, Sommer A, Raposo do Amaral CM, Gorlin RJ, Mulliken JB, Olsen BR. Autosomal dominant craniometaphyseal dysplasia is caused by mutations in the transmembrane protein ANK. Am J Hum Genet. 2001 Jun;68(6):1321-6. doi: 10.1086/320612. Epub 2001 Apr 16. PMID 11326338
- [Result] Hu Y, Chen IP, de Almeida S, Tiziani V, Do Amaral CM, Gowrishankar K, Passos-Bueno MR, Reichenberger EJ. A novel autosomal recessive GJA1 missense mutation linked to Craniometaphyseal dysplasia. PLoS One. 2013 Aug 12;8(8):e73576. doi: 10.1371/journal.pone.0073576. eCollection 2013. PMID 23951358
- [Result] Dutra EH, Chen IP, Reichenberger EJ. Dental abnormalities in a mouse model for craniometaphyseal dysplasia. J Dent Res. 2013 Feb;92(2):173-9. doi: 10.1177/0022034512468157. Epub 2012 Nov 15. PMID 23160629
- [Result] Chen IP, Tadinada A, Dutra EH, Utreja A, Uribe F, Reichenberger EJ. Dental Anomalies Associated with Craniometaphyseal Dysplasia. J Dent Res. 2014 Jun;93(6):553-8. doi: 10.1177/0022034514529304. Epub 2014 Mar 24. PMID 24663682
- [Result] Chen IP, Luxmi R, Kanaujiya J, Hao Z, Reichenberger EJ. Craniometaphyseal Dysplasia Mutations in ANKH Negatively Affect Human Induced Pluripotent Stem Cell Differentiation into Osteoclasts. Stem Cell Reports. 2017 Nov 14;9(5):1369-1376. doi: 10.1016/j.stemcr.2017.09.016. Epub 2017 Oct 19. PMID 29056330
- [Result] Kanaujiya J, Bastow E, Luxmi R, Hao Z, Zattas D, Hochstrasser M, Reichenberger EJ, Chen IP. Rapid degradation of progressive ankylosis protein (ANKH) in craniometaphyseal dysplasia. Sci Rep. 2018 Oct 24;8(1):15710. doi: 10.1038/s41598-018-34157-5. PMID 30356088
- [Result] Fujii Y, Kozak E, Dutra E, Varadi A, Reichenberger EJ, Chen IP. Restriction of Dietary Phosphate Ameliorates Skeletal Abnormalities in a Mouse Model for Craniometaphyseal Dysplasia. J Bone Miner Res. 2020 Oct;35(10):2070-2081. doi: 10.1002/jbmr.4110. Epub 2020 Jul 12. PMID 33463757
- See also: study website — https://health.uconn.edu/reichenberger-lab/